CLINICAL TRIAL: NCT05132491
Title: Evaluation of a Technology Early Career Preparation Intervention (TECH-Prep) for African American Young Adults With Developmental Disabilities
Brief Title: Benefits of Coding Training on Young Adults With Developmental Disabilities
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0842; A177800 (Other: UW Madison); EDUC/REHAB PSYCH & SPEC ED (Other: UW Madison); FP00010584_SA003 (Other Grant/Funding Number: DHHS)
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Developmental Disability
Keywords: STEM; Career Interest; underserved populations; education
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online Training Program (Experimental): An online intervention for people with disabilities intended to increase social skills and interest in coding careers.
  Interventions: Other: TECH-Prep Intervention

INTERVENTIONS:
Other: TECH-Prep Intervention — Participants in the treatment program will be asked to complete 10 online training modules (1 hour each), attend 5 online motivational speaker forums (1 hour each), and view 5 coding workshops. The activities will be completed over an 8 week period.

SUMMARY:
The purpose of the present study is to develop and evaluate the Technology Early Career Preparation Intervention (TECH-Prep) program with African American high school students with developmental disabilities. Developmental disabilities include conditions such as Autism spectrum disorders, seizure disorders, behavior disorders, brain injury, cerebral palsy, Down syndrome, and fetal alcohol syndrome/effects. This program is designed to increase technology career interests, self-efficacy, outcome expectancy, goal persistence, and increase entrance into post-secondary education or work subsequent to high school completion of African American youth with developmental disabilities.

DETAILED DESCRIPTION:
The investigator's goal is to recruit 30 African American high school students with developmental disabilities to participate in this TECH-Prep study each year for the next five years (2019-2024). The TECH-Prep program integrates many empirically supported strategies identified in the STEM education and the secondary transition research literature. The program will incorporate overview of coding careers, reviewing video testimonials of individuals working in technology fields, and reviewing/responding to training materials intended to facilitate workplace social skills development.

The program will require participants complete three surveys to track their progress. To receive incentives for completing program components, data on program component completion will be tracked of participants in the treatment group. This involves tracking data on when a participant completes review of the final segment of each learning module.

Data collection for this study will consist of three surveys completed at baseline, immediately after completion of the program, and six weeks after completion of the program.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of diverse racial and cultural backgrounds
* Diagnosed with a developmental disability
* Over 18 but under 24
* Have the capacity to provide informed consent

Exclusion Criteria:

* Persons who are Caucasian
* Do not have a developmental disability
* Older than 24 years of age
* Unable to provide informed consent

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in Outcome Expectation Sub-score on the Tech-Prep Survey | baseline, 2 weeks (immediately after intervention), 8 weeks (6 weeks post intervention)
  The Tech-Prep survey is a 90-item survey. Scores are calculated on sub-scales included in the survey. These subscales focus on Social Cognitive Career Theory concepts of outcome expectation, career readiness, and goal persistence. Change scores from baseline at post-training and post-internship will be evaluated. Higher scores indicate increased outcome expectations.
Change in Goal Persistence Sub-score on the Tech-Prep Survey | baseline, 2 weeks (immediately after intervention), 8 weeks (6 weeks post intervention)
  The Tech-Prep survey is a 90-item survey. Scores are calculated on sub-scales included in the survey. These subscales focus on Social Cognitive Career Theory concepts of outcome expectation, career readiness, and goal persistence. Change scores from baseline at post-training and post-internship will be evaluated. Higher scores indicate increased goal persistence.
Change in Career Readiness Sub-score on the Tech-Prep Survey | baseline, 2 weeks (immediately after intervention), 8 weeks (6 weeks post intervention)
  : The Tech-Prep survey is a 90-item survey. Scores are calculated on sub-scales included in the survey. These subscales focus on Social Cognitive Career Theory concepts of outcome expectation, career readiness, and goal persistence. Change scores from baseline at post-training and post-internship will be evaluated. Higher scores indicate increased career readiness.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Tansey, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No